CLINICAL TRIAL: NCT07250217
Title: Collection of Biological Samples for Research Purposes: Determination of Epigenetic Markers of Acute Myeloblastic Leukemia in Elderly Patients
Brief Title: Determination of Epigenetic Markers of Acute Myeloblastic Leukemia in Elderly Patients
Acronym: LAMME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Collaborators: Institut de Recherche en Hématologie et Transplantation (IRHT) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GHRMSA 1447
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloblastic Leukemia
Keywords: Acute Myeloblastic Leukemia; Methylome; Epigenetic markers; Bone marrow; Diagnosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AML (Other): Elderly patients diagnosed with acute myeloid leukemia. An additional volume of blood (10 mL) and bone marrow (2 mL) will be collected during follow-up visits as part of their routine care.
  Interventions: Diagnostic Test: Epigenetic markers
- Control group (Other): Elderly patients scheduled for thoracic surgery involving sternotomy. A bone marrow sample (2 mL) will be obtained by sternal puncture in the operating room (after general anesthesia and before sternotomy), and an additional blood sample (10 mL) will be collected during the hospital stay.
  Interventions: Diagnostic Test: Epigenetic markers

INTERVENTIONS:
Diagnostic Test: Epigenetic markers — Methylation profiles will be analyzed and DNA regions (CpG sites) that show significant differences between healthy and pathological cells from bone marrow will be identified. These regions could serve as epigenetic markers for cells from patients with LAM, if they can be used by digital PCR. These differentially methylated CpG islands will be targeted for the design of specific primer and probe pairs for use in digital PCR. The markers will then be tested in circulating free DNA from blood.

SUMMARY:
The main objective of this study is to identify epigenetic markers specific to abnormal myeloid cells in patients with acute myeloid leukemia (AML) by analyzing the methylation of circulating cell-free DNA in plasma.

DETAILED DESCRIPTION:
Secondary objectives:

* To evaluate the correlation between epigenetic markers and clinical response to treatment with Azacytidine.
* To compare methylation patterns between patients who respond and those who do not respond to treatment of AML.

Conduct of research:

This study will allow the collection of samples for the establishment of a biobank. The study population is divided into two groups:

Control group: Elderly patients scheduled for thoracic surgery involving sternotomy. A bone marrow sample (2 mL) will be obtained by sternal puncture in the operating room (after general anesthesia and before sternotomy), and an additional blood sample (10 mL) will be collected during the hospital stay.

AML group: Elderly patients diagnosed with acute myeloid leukemia. An additional volume of blood (10 mL) and bone marrow (2 mL) will be collected during follow-up visits as part of their routine care.

ELIGIBILITY:
1. / Control Group

   Inclusion Criteria:
   * Age ≥ 60 years;
   * Scheduled for cardiac surgery involving sternotomy;
   * Normal blood count within the two months preceding sampling;
   * Affiliated with, or beneficiary of, a social security system;
   * Written informed consent to participate in the study.

   Exclusion Criteria:
   * Patients deemed unsuitable for sampling by the surgeon performing the procedure;
   * Patients under legal protection measures;
   * Patients under judicial supervision or deprived of liberty by judicial or administrative decision;
   * Presence of positive virological markers indicating active infection (hepatitis B, hepatitis C, or HIV).
2. / AML Group

Inclusion Criteria:

* Age ≥ 60 years;
* Diagnosis of de novo AML or AML secondary to myelodysplastic syndrome, scheduled to receive azacitidine-based treatment;
* Affiliated with, or beneficiary of, a social security system;
* Written informed consent to participate in the study.

Exclusion Criteria:

* Diagnosis of a hematologic disease other than AML;
* Clinical signs suggestive of active central nervous system leukemia, or presence of isolated extramedullary leukemia;
* Previous treatment for AML other than hydroxyurea;
* Severe comorbidities that could interfere with the study, as assessed by the principal investigator;
* Presence of positive virological markers indicating active infection (hepatitis B, hepatitis C, or HIV);
* Patients under legal protection;
* Patients under judicial supervision or deprived of liberty by judicial or administrative decision.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of methylation of specific CpG sites | Baseline
  The methylation of circulating free DNA in plasma is quantified by measuring the percentage of methylation of specific CpG motifs analyzed in cfDNA relative to total methylation.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Groupe Hospitalier de la Région de Mulhouse et Sud Alsace, Mulhouse, Alsace
  - GHRMSA, Mulhouse

IPD SHARING:
Plan to Share IPD: No